CLINICAL TRIAL: NCT05161260
Title: Pilot Study of Group Video Yogic Breathing App in Breast Cancer Survivors
Brief Title: Breathwork App for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sundar Balasubramanian (Industry)
Collaborators: PranaScience Institute LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sundar Balasubramanian, Principal Investigator, Founder, Owner, PranaScience Institute LLC
Organization: PranaScience Institute LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 108511; 1R41CA254557-01A1 (NIH); R41CA254557 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2021-12-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Breathing (YB) (Experimental): A first production version of a mobile application that guides users through proscribed yoga breathing exercises.
  Interventions: Behavioral: Yoga Breathing
- Attention Control (Experimental): A first production version of a mobile application that guides users through an attention control activity, presented as methods for mindfulness.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Yoga Breathing — For the12 weeks, participants will be asked to use the mobile study app, completing 3, 10 minute exercises, 5 days a week. Participants in the Yoga Breathing group will practice a breathing exercise guided by the mobile study application. The application will also send "nudges" and reminders throughout the day. Participants will engage with the research study app along with other participants in groups of 2-7 at their own convenience. Participants may practice their breathing activity with either a group of participants, through the video conferencing feature of the app, or on their own. The study instructor may join sessions on a random basis to ensure compliance with the technique and to clarify any questions participants may have.
  Other Names: YB
  Arms: Yoga Breathing (YB)
Behavioral: Attention Control — For the12 weeks, participants will be asked to use the mobile study app, completing 3, 10 minute exercises, 5 days a week. Participants in the Attention Control group will practice a mindfulness exercise guided by the mobile study application. The application will also send "nudges" and reminders throughout the day. Participants will engage with the research study app along with other participants in groups of 2-7 at their own convenience. Participants may practice their mindfulness activity with either a group of participants, through the video conferencing feature of the app, or on their own. The study instructor may join sessions on a random basis to ensure compliance with the technique and to clarify any questions participants may have.
  Other Names: Mindfulness
  Arms: Attention Control

SUMMARY:
Cancer survivorship is associated with many long-term chronic health issues that arise as a result of cancer treatment protocols. Non-pharmacological lifestyle and mind-body interventions have been shown to be effective and critical components of a total-health strategy for cancer survivors. PranaScience Institute seeks to develop and test a novel group video app for home-based delivery of a Yogic Breathing intervention that reduces symptoms of cancer treatment survival and supports total-health.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, willing to provide informed consent.
2. Diagnosis of Stage 0-III breast cancer.
3. Completion of radiation therapy within the last 6 months.
4. ECOG performance status of 0-3 during cancer treatment.
5. Orally expressed visual and auditory acuity adequate for filling out all study forms and participating in telephone interviews and internet-based group video applications.
6. Access to telephone and internet-connected computer or mobile phone.

Exclusion Criteria:

1. Subject is unwilling or unable to comply with any of the study procedures.
2. Orally expressed dependence on alcohol or drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Total practice time as assessed in minutes within the study application. | 12 weeks
  Adherence will be evaluated by assessing total practice times by length in minutes.
Total practice time as assessed in frequency of using the study application. | 12 weeks
  Adherence will be evaluated by assessing total practice times by total number of times per day using the application.
Participants' symptom management as measured by emotional disposition. | 12 weeks
  Acceptability measures the participant's symptom management throughout the study duration. Participant's emotional disposition at the beginning and end of each study session with the Smiley Face Likert Scale, exhibiting as Very Poor, Poor, Average, Good, or Excellent to measure participants' acceptability of the study application.
Participants' symptom management as measured by the System Usability Scale. | 12 weeks
  Acceptability measures the participant's symptom management throughout the study duration. This is measured using The System Usability Scale (SUS) questionnaire, a 10 item questionnaire with 5 response options ranging from 'Strong Agree' to 'Strong Disagree'. The questionnaire will be administered at the end of 12 weeks to measure participants' acceptability of the study application.
Participants' symptom management as measured by a focus group. | 12 weeks
  Acceptability measures the participant's symptom management throughout the study duration. Input from end of study Focus Groups will be used to measure participants' acceptability of the study application.
Feasibility of study application measured by participant ability to perform all study procedures. | 12 weeks
  Feasibility for use of study application will be measured by evaluating intervention delivery factors, which will be evaluated throughout the program period by examining the total number of participants who completed all study sessions.

SECONDARY OUTCOMES:
Behavioral Survey Measures through Perceived Stress. | 12 weeks
  Behavioral survey measures will be collected from all participants at study start and study termination using established questionnaires: Perceived Stress Scale (PSS), a 10 item questionnaire with 5 response options ranging from 'Never' to 'Very Often', with 'Very Often' being a worse outcome.
Behavioral Survey Measures through Depression Scale. | 12 weeks
  Behavioral survey measures will be collected from all participants at study start and study termination using established questionnaires: Depression Scale, a questionnaire with 4 response options ranging from 'Not at all' to 'Most of the time', with 'Most of the time' being a worse outcome.
Behavioral Survey Measures through MD Anderson Symptom Inventory. | 12 weeks
  Behavioral survey measures will be collected from all participants at study start and study termination using established questionnaires: MD Anderson Symptom Inventory, a 13 symptom list with responses on a scale of 0 to 10, with 10 being the worst outcome.
Study participant focus group interviews. | 16 weeks
  Structured focus group interviews completed approximately 1 month after the end of the 12 week intervention. This will assess participants' general perceptions of the intervention and technology. During these interviews, data will be collected to identify recommendations for app modifications and improved adherence.
Exploratory salivary biomarkers to indicate changes. | 12 weeks
  Participants will each be asked to provide a total of 8 saliva samples (1 pre and post study session at Week 1 and Week 12). Proteomic, multiplex, and ELISA will be used to measure changes in cytokines, tumor suppressors, and cortisol.
Exploratory fingernail biomarkers to indicate changes. | 12 weeks
  Participants will each be asked to provide a total of 16 fingernail samples (8 at Week 1 and 8 at Week 12). Proteomic, multiplex, and ELISA will be used to measure changes in cytokines, tumor suppressors, and cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Balasubramanian, PhD, Principal Investigator — PranaScience; Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: : Individual participant data requests can be submitted starting 9 months after research article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: "Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the PI.

REFERENCES:
- [Derived] Balasubramanian S, Harper J, Sterba KR, Viswanathan R, Eldredge-Hindy H. Protocol for the Pilot Study of Group Video Yogic Breathing App in Breast Cancer Survivors. Int J Aayush Tradit Med. 2022;2(2):38-57. Epub 2022 Sep 28. PMID 36790946